CLINICAL TRIAL: NCT06396793
Title: Prevalence of Psychological Symptoms and Their Correlation With the Rehabilitative Outcome in Patients With Cardiac and Pulmonary Diseases Undergoing a Hospital Rehabilitation.
Brief Title: Psychological Symptoms in Cardiac and Pulmonary Diseases
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Other Study IDs: CEC N. 2695
Record Dates: First submitted 2024-04-30; First posted 2024-05-02 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Psychological Distress; Anxiety; Depression; Cardiovascular Diseases; Pulmonary Disease; Rehabilitation; Coping Behavior
MeSH Terms: conditions — Anxiety Disorders; Depression; Cardiovascular Diseases; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardio-respiratory: Inpatients affected by cardiac or pulmonary diseases undergoing a rehabilitative program
  Interventions: Other: no intervention because it is an observational study

INTERVENTIONS:
Other: no intervention because it is an observational study — it is an observational study thus there is no intervention

SUMMARY:
The European guidelines emphasize the importance of conducting psychological screenings to investigate the presence of stress and symptoms of anxiety and depression in patients with cardiovascular disease: depression, common among patients with CVD, is associated with increased mortality, disability, decreased adherence to healthy lifestyles and medical treatments, and together with anxiety, the risk of mortality increases by about 3 times; stress, furthermore, is associated with the development and progression of cardiovascular diseases and is correlated with low adherence and cigarette smoking.

Less studied, but not less important, are the incidence of anxiety, depression, and stress in pulmonary disease, the relationship between mental disorders and pulmonary diseases, as well as the effect of the psychological component on the rehabilitative outcome of such patients: for example, there is evidence that those suffering from chronic obstructive pulmonary disease (COPD) present symptoms of depression and anxiety much more frequently than the general population and that these two mental disorders may exacerbate COPD itself.

The literature, therefore, highlights that the risk of onset of cardiovascular disease increases with the severity of mental disorder, and some psychological variables correlate with the outcomes of cardiac rehabilitation intervention, crucial for reducing rehospitalizations, myocardial infarction, and mortality, as well as for improving the patient's quality of life and ability to perform physical exercises.

In light of this evidence and the recent recommendations of the ESC, the present study aims to conduct screening for symptoms of anxiety, depression, and stress in all patients admitted to the Cardiology and Pulmonary Rehabilitation Units of the Milan Center, Camaldoli in order to assess their incidence and to select, through validated tools, patients who require personalized psychological intervention based on their level of risk, correlating then the presence of such symptoms with the rehabilitative outcome, in order to assess how much the mental component interferes with the care pathway. The level of acceptance and feasibility of a computerized data collection procedure will also be evaluated, a procedure that, if well accepted, would make the screening process much simpler, safer, and more economical.

ELIGIBILITY:
Inclusion Criteria:

* aged≥18
* able to fulfil questionnaires autonomously

Exclusion Criteria:

* no Italian comprehension,
* severe visuoperceptive deficits,
* cognitive deterioration preventing self-completion of questionnaires,
* refusal to underwent to the evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the ICS Maugeri Cardiology and Pulmonary Rehabilitation Units
Sampling Method: Non-Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of psychological risk and protective factors | 18 months
  To conduct a screening of anxious, depressive, stress symptoms and coping strategies in patients admitted a Cardiology and pulmonary Rehabilitation Units

SECONDARY OUTCOMES:
Correlations between psychological variables and rehabilitative outcomes | 18 months
  To correlate risk and protective factors with rehabilitative outcomes
Acceptance of computerized screening | 18 months
  The degree of acceptance of an online data collection procedure will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Gorini, PhD, Principal Investigator — ICS Maugeri SpA SB
Locations (1):
- ICS Maugeri SpA SB, Milan, MI, Italy

REFERENCES:
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC National Cardiac Societies; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur Heart J. 2021 Sep 7;42(34):3227-3337. doi: 10.1093/eurheartj/ehab484. No abstract available. PMID 34458905
- [Background] Celano CM, Suarez L, Mastromauro C, Januzzi JL, Huffman JC. Feasibility and utility of screening for depression and anxiety disorders in patients with cardiovascular disease. Circ Cardiovasc Qual Outcomes. 2013 Jul;6(4):498-504. doi: 10.1161/CIRCOUTCOMES.111.000049. Epub 2013 Jun 11. PMID 23759474
- [Background] MacGregor KL, Funderburk JS, Pigeon W, Maisto SA. Evaluation of the PHQ-9 Item 3 as a screen for sleep disturbance in primary care. J Gen Intern Med. 2012 Mar;27(3):339-44. doi: 10.1007/s11606-011-1884-5. Epub 2011 Sep 24. PMID 21948205
- [Background] Vaccarino V, Badimon L, Bremner JD, Cenko E, Cubedo J, Dorobantu M, Duncker DJ, Koller A, Manfrini O, Milicic D, Padro T, Pries AR, Quyyumi AA, Tousoulis D, Trifunovic D, Vasiljevic Z, de Wit C, Bugiardini R; ESC Scientific Document Group Reviewers. Depression and coronary heart disease: 2018 position paper of the ESC working group on coronary pathophysiology and microcirculation. Eur Heart J. 2020 May 1;41(17):1687-1696. doi: 10.1093/eurheartj/ehy913. No abstract available. PMID 30698764
- [Background] Reavell J, Hopkinson M, Clarkesmith D, Lane DA. Effectiveness of Cognitive Behavioral Therapy for Depression and Anxiety in Patients With Cardiovascular Disease: A Systematic Review and Meta-Analysis. Psychosom Med. 2018 Oct;80(8):742-753. doi: 10.1097/PSY.0000000000000626. PMID 30281027
- [Background] Crawshaw J, Auyeung V, Norton S, Weinman J. Identifying psychosocial predictors of medication non-adherence following acute coronary syndrome: A systematic review and meta-analysis. J Psychosom Res. 2016 Nov;90:10-32. doi: 10.1016/j.jpsychores.2016.09.003. Epub 2016 Sep 8. PMID 27772555
- [Background] Maurer J, Rebbapragada V, Borson S, Goldstein R, Kunik ME, Yohannes AM, Hanania NA; ACCP Workshop Panel on Anxiety and Depression in COPD. Anxiety and depression in COPD: current understanding, unanswered questions, and research needs. Chest. 2008 Oct;134(4 Suppl):43S-56S. doi: 10.1378/chest.08-0342. PMID 18842932
- [Background] Anderson L, Oldridge N, Thompson DR, Zwisler AD, Rees K, Martin N, Taylor RS. Exercise-Based Cardiac Rehabilitation for Coronary Heart Disease: Cochrane Systematic Review and Meta-Analysis. J Am Coll Cardiol. 2016 Jan 5;67(1):1-12. doi: 10.1016/j.jacc.2015.10.044. PMID 26764059
- [Background] Salzwedel A, Jensen K, Rauch B, Doherty P, Metzendorf MI, Hackbusch M, Voller H, Schmid JP, Davos CH. Effectiveness of comprehensive cardiac rehabilitation in coronary artery disease patients treated according to contemporary evidence based medicine: Update of the Cardiac Rehabilitation Outcome Study (CROS-II). Eur J Prev Cardiol. 2020 Nov;27(16):1756-1774. doi: 10.1177/2047487320905719. Epub 2020 Feb 23. PMID 32089005
- [Background] Taylor RS, Walker S, Smart NA, Piepoli MF, Warren FC, Ciani O, Whellan D, O'Connor C, Keteyian SJ, Coats A, Davos CH, Dalal HM, Dracup K, Evangelista LS, Jolly K, Myers J, Nilsson BB, Passino C, Witham MD, Yeh GY; ExTraMATCH II Collaboration. Impact of Exercise Rehabilitation on Exercise Capacity and Quality-of-Life in Heart Failure: Individual Participant Meta-Analysis. J Am Coll Cardiol. 2019 Apr 2;73(12):1430-1443. doi: 10.1016/j.jacc.2018.12.072. PMID 30922474
- [Background] Long L, Mordi IR, Bridges C, Sagar VA, Davies EJ, Coats AJ, Dalal H, Rees K, Singh SJ, Taylor RS. Exercise-based cardiac rehabilitation for adults with heart failure. Cochrane Database Syst Rev. 2019 Jan 29;1(1):CD003331. doi: 10.1002/14651858.CD003331.pub5. PMID 30695817